CLINICAL TRIAL: NCT03873974
Title: Multicentre Clinical Trial to Assess the Performance of the DualDur In Vitro Diagnostic System in the Diagnosis of Lyme Borreliosis From Blood Samples of Subjects Who Are Either Pharmacotherapy-naive or Treatment-experienced and Their Physician Indicates Drug Therapy for Lyme Borreliosis
Brief Title: Performance Evaluation of the DualDur In Vitro Diagnostic System in the Diagnosis of Lyme Borreliosis
Status: Completed | Type: Observational
Sponsor: Lyme Diagnostics Ltd. (Industry)
Collaborators: Pharmahungary Group (Industry)
Responsible Party: Sponsor
Other Study IDs: LymeDD_CIP
Record Dates: First submitted 2019-02-28; First posted 2019-03-14 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-01

CONDITIONS: Lyme Borreliosis
Keywords: Lyme Borreliosis; Lyme disease; In Vitro Diagnostics System; Dark Field Microscopy
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples will be collected from patients and healthy volunteers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Negative trial arm: Venous blood samples will be taken for central laboratory analysis with:
  * DualDur dark-field microscopic test
  * DualDur dark-field automatic microscopic test
  * Western blot IgM and IgG
  * Bózsik Western blot IgM and IgG
  * Enzyme-Linked Immunosorbent Assay (ELISA) IgM and IgG
  * DualDur Polymerase chain reaction
  Interventions: Diagnostic Test: DualDur dark-field microscopic test; Diagnostic Test: DualDur dark-field automatic microscopic test; Diagnostic Test: Western blot IgM and IgG; Diagnostic Test: Bózsik Western blot IgM and IgG; Diagnostic Test: enzyme-linked immunosorbent assay (ELISA) IgM and IgG; Diagnostic Test: DualDur Polymerase chain reaction
- Positive trial arm: Venous blood samples will be taken for central laboratory analysis with:
  * DualDur dark-field microscopic test
  * DualDur dark-field automatic microscopic test
  * Western blot IgM and IgG
  * Bózsik Western blot IgM and IgG
  * Enzyme-Linked Immunosorbent Assay (ELISA) IgM and IgG
  * DualDur Polymerase chain reaction
  Interventions: Diagnostic Test: DualDur dark-field microscopic test; Diagnostic Test: DualDur dark-field automatic microscopic test; Diagnostic Test: Western blot IgM and IgG; Diagnostic Test: Bózsik Western blot IgM and IgG; Diagnostic Test: enzyme-linked immunosorbent assay (ELISA) IgM and IgG; Diagnostic Test: DualDur Polymerase chain reaction

INTERVENTIONS:
Diagnostic Test: DualDur dark-field microscopic test — Morphologically identify the presence of Borrelia burgdorferi sensu lato bacteria (in a broader sense) which are present in the body fluid, hence to verify Borreliosis. Manual evaluation.
Diagnostic Test: DualDur dark-field automatic microscopic test — Morphologically identify the presence of Borrelia burgdorferi sensu lato bacteria (in a broader sense) which are present in the body fluid, hence to verify Borreliosis. Software evaluation.
Diagnostic Test: Western blot IgM and IgG — Borrelia qualitative in vitro test in order to detect and reliably identify IgG and IgM antibodies against Borrelia burgdorferi from human serum or plasma.
Diagnostic Test: Bózsik Western blot IgM and IgG — Borrelia qualitative in vitro test in order to detect and reliably identify IgG and IgM antibodies against Borrelia burgdorferi from human serum or plasma.
Diagnostic Test: enzyme-linked immunosorbent assay (ELISA) IgM and IgG — Standard ELISA test for Lyme borreliosis.
Diagnostic Test: DualDur Polymerase chain reaction — DualDur PCR test for Lyme borreliosis.

SUMMARY:
The clinical data from the clinical trial will be used to assess the performance, sensitivity and specificity of the experimental DualDur In Vitro Diagnostic System.

DETAILED DESCRIPTION:
The clinical data from the clinical trial will be used to assess the performance, sensitivity and specificity of the experimental DualDur In Vitro Diagnostic System.

* The sensitivity of the DualDur in Vitro Diagnostic System will be examined in subjects whose physician indicates drug therapy for Lyme borreliosis (positive arm).
* The specificity of the DualDur in Vitro Diagnostic System will be examined in healthy volunteers declared Lyme borreliosis negative by their physician and all the standard laboratory tests prove that they are free of Lyme borreliosis (negative arm).

The diagnostic system developed by Lyme Diagnostics Ltd. is planned for application in the diagnosis during the entire life cycle of Lyme borreliosis.

ELIGIBILITY:
I. Positive trial arm

I.1. Inclusion Criteria:

* Man or female subjects over 18 years of age
* Treatment-naive or treatment-experienced subjects with Lyme borreliosis, whose physician indicates drug therapy for Lyme borreliosis.
* Subjects capable of reading, understanding, and observing the requirements of the clinical trial, who sign the Patient Information Leaflet and Informed Consent Form approved by the Competent Authority and the Ethics Committee.

I. 2. Exclusion Criteria:

* Man or female subjects over 80 years of age
* Pregnancy, breastfeeding
* History of any complication related to previous blood sampling
* Coagulation and/or bleeding disorders
* Anticoagulant therapy
* Acute, life-threatening condition
* Participation in another clinical trial
* The patient is under antibiotic therapy, or received such treatment in the preceding 3 months
* The patient is currently taking or has taken in the preceding 6 months dietary supplements of herbal origin, or medicinal herbs as first-line or add-on treatments for Lyme borreliosis
* In the event the patient has previously been treated for Lyme borreliosis, then this treatment took place less than 6 months before blood sampling.
* In the preceding 6 months, the patient used an electronic device operating along the principle of electromagnetic (i.e. electric or magnetic) fields - such as bioresonance, pulsed magnetic field, etc. - as add-on treatment for Lyme borreliosis.

II. Negative trial arm

II.1. Inclusion Criteria:

* Man or female subjects over 18 years of age
* Asymptomatic healthy volunteer subjects without acute or chronic symptoms of Lyme borreliosis, who are free of Lyme borreliosis by the indication of all standard laboratory tests, and who are willing to take part in a comprehensive medical examination and related blood sampling.
* Subjects capable of reading, understanding, and observing the requirements of the trial, who sign the Patient Information Leaflet and Informed Consent Form approved by the Competent Authority and the Ethics Committee.

II. 2. Exclusion Criteria:

* Man or female subjects over 80 years of age
* Pregnancy, breastfeeding
* History of any complication related to previous blood sampling
* Coagulation and/or bleeding disorders
* Anticoagulant therapy
* Participation in another clinical trial
* Lyme borreliosis diagnosed previously, at any time during the life of the subject
* The subject has received any treatment for Lyme borreliosis (medicinal products, dietary supplements, medicinal plants, electronic devices, etc.) during his/her life
* The patient is under antibiotic therapy, or received such treatment in the preceding 3 months
* The occupation of the subject is either a forester or a hunter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Positive trial arm: At least 18-year-old, treatment-naive or treatment-experienced men and women with Lyme borreliosis, whose physician indicates drug therapy for Lyme borreliosis. Furthermore, they consent to the collection and processing of their data during the clinical trial, and to blood sampling for the assessment of the DualDur IVD System, and to the diagnostic analyses of these samples in the central laboratory of the trial.
  Negative trial arm: At least 18-year-old healthy volunteers without the symptoms of either acute or chronic Lyme borreliosis, who have not been treated for Lyme borreliosis, and all the standard laboratory tests prove that they are free of Lyme borreliosis.
  Furthermore, they give their consent to blood sampling for the purposes of the clinical trial, to the collection and processing of their data, and to the analyses of their blood samples in the central laboratory of the trial.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Primary endpoint, 1 (sensitivity of the experimental DualDur in Vitro Diagnostic System) | Laboratory samples evaluated within 72-144 hours of sampling.
  The sensitivity of the experimental DualDur in Vitro Diagnostic System in the positive arm, based on medical diagnosis
Primary endpoint, 2 (specificity of the experimental DualDur In Vitro Diagnostic System) | Laboratory samples evaluated within 72-144 hours of sampling.
  The specificity of the experimental DualDur In Vitro Diagnostic System in the negative arm, based on medical diagnosis and all the standard laboratory test results

SECONDARY OUTCOMES:
Secondary endpoint, 1 (sensitivity of the experimental DualDur in Vitro Diagnostic System) | Laboratory samples evaluated within 72-144 hours of sampling.
  1. The sensitivity of the experimental DualDur in Vitro Diagnostic System, based on medical diagnosis (Lyme borreliosis positive) and direct/indirect diagnostic methods.
Secondary endpoint, 2 (Pairwise comparison of the sensitivity of the experimental DualDur in Vitro Diagnostic System and of the direct/indirect diagnostic methods) | Laboratory samples evaluated within 72-144 hours of sampling.
  Pairwise comparison of the sensitivity of the experimental DualDur in Vitro Diagnostic System and of the direct/indirect diagnostic methods

OTHER OUTCOMES:
Tertiary endpoint (Validation of the image evaluation) | Software evaluation done at planned study completion date, February 2020.
  Validation of the image evaluation software applied in the diagnosis of Lyme borreliosis by dark field microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Bela P. Bozsik, MD, Study Director — Lyme Diagnostics Ltd.
Locations (8):
- MedUni Vienna,University Hospital Internal Medicine I, Clinical Dept. for Infections, Vienna, Austria
- Czechia (2):
  - FORBELI s.r.o., Prague
  - Neurologická ambulance, Prague
- Praxis Dr.med. Reinhardt, Pforzheim, Germany
- Istenhegyi Géndiagnosztika Magánorvosi Rendelő Ltd., Budapest, Hungary
- Poland (2):
  - St. Luke's Clinic, Gdansk
  - Centrum Dr. Ozimek, Warsaw
- Borélia centrum Bratislava, BCB Clinic, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided
To be decided later.

REFERENCES:
- See also: Official website of study Sponsor, Lyme Diagnostics Ltd. — http://lymediagnostics.com/
- See also: Official website of central laboratory, Synlab Hungary Ltd. — https://www.synlab.hu/
- See also: European Parliament Resolution of 15 November 2018 on Lyme disease (Borreliosis) (2018/2774(RSP) — http://www.europarl.europa.eu/sides/getDoc.do?pubRef=-//EP//NONSGML+TA+P8-TA-2018-0465+0+DOC+PDF+V0//EN
- See also: Official website of CRO, Pharmahungary Group. — http://www.pharmahungary.com/